CLINICAL TRIAL: NCT03252522
Title: Evaluating the Efficacy of Supplementation With Micronutrients for ADHD in Youth (MADDY) Study
Brief Title: Micronutrients for Attention-Deficit Hyperactivity Disorder in Youth (MADDY) Study
Acronym: MADDY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Ohio State University (Other); University of Lethbridge (Other); National University of Natural Medicine (Other); Foundation for Excellence in Mental Health Care (Other); The Waterloo Foundation (Other)
Responsible Party: Principal Investigator, Jeanette Johnstone, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16870
Record Dates: First submitted 2017-07-26; First posted 2017-08-17 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; ODD; DMDD; Inattention; Impulsivity; Irritability; Anger; Micronutrients; Emotional Dysregulation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Impulsive Behavior | interventions — Minerals; Amino Acids; Antioxidants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo-controlled; randomization created by statistician, all involved in the study and assessment are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Capsules of broad spectrum micronutrients: a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants.
  Interventions: Combination Product: Broad Spectrum Micronutrients; a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants
- Placebo (Placebo Comparator): Capsules of inactive placebo.
  Interventions: Dietary Supplement: Placebo
- Open Label (Experimental): All participants have the option to participate in an 8-week, naturalistic, open label follow-up in which the child will take the active micronutrient treatment; capsules of broad spectrum micronutrients.
  Interventions: Combination Product: Broad Spectrum Micronutrients; a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants

INTERVENTIONS:
Combination Product: Broad Spectrum Micronutrients; a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants — 60% of participants will take 3-4 capsules of broad spectrum micronutrients three times per day for eight weeks. Following the initial 8 weeks (of the RCT), all participants will have the option to participate in an open label extension, during which time the child would take the active micronutrient treatment for 8 weeks
  Other Names: Daily Essential Nutrients (DEN)
  Arms: Intervention; Open Label
Dietary Supplement: Placebo — 40% of participants will take 3-4 capsules of inactive placebo three times per day for eight weeks.
  Arms: Placebo

SUMMARY:
This proposed research will use randomized control trial (RCT) methodology and compare micronutrients with placebo in 135 children with ADHD.

DETAILED DESCRIPTION:
This study examines a broad spectrum micronutrient treatment for children with ADHD. The goal is to broaden the scope of evidence-based treatments, and to address the public desire for non-pharmacological treatment options. This study will use a randomized controlled trial design, comparing micronutrients with placebo in 135 children, ages 6-12, with ADHD plus irritability or anger based on parent-report of symptoms. The study will also collect biological samples (saliva, stool, urine, hair, and blood) from the children to examine physiological mechanisms of micronutrient effects. If the micronutrient treatment successfully diminishes symptoms, the clinical implication is to offer this as a legitimate non-pharmacological alternative to stimulant medication.

ELIGIBILITY:
Inclusion Criteria:

* Age inclusive of and between 6 and 12 years at the time of enrollment.
* Verbally willing to swallowing a maximum of 9-12 capsules/day with food, attend all study appointments and complete questionnaires.
* Meet criteria for ADHD as assessed by the clinical cut-off (6+ questions scored as 2's or 3's, "often," or "very often") on the Category A: ADHD questions from on the Child & Adolescent Symptom Inventory-5 (CASI-5) with at least several symptoms present in more than one setting, based on the Diagnostic and Statistical Manual (DSM) 5 symptom criteria, including significant impairment in functioning socially and/or academically.
* Demonstrate at least one symptom of irritability or anger as assessed by a score of 2 or 3 on one question from Category B or Rz from the CASI-5.
* Be medication-free, or washout with medical supervision to be provided by the child's pediatrician or primary care physician, reliant on the parent/guardian to work with that physician, for at least two weeks prior to in-person study assessment. Washout will be recorded as occurring on the date reported by the parent/guardian, with a faxed copy of the progress note, visit summary or signed letter from participant's doctor.

Exclusion Criteria:

* Neurological disorder involving brain or other central function (e.g., history of or suspected intellectual disability, autism spectrum disorder, epilepsy, multiple sclerosis, narcolepsy) or other major psychiatric condition requiring hospitalization (e.g. significant mood disorder, active suicidal ideation, or psychosis), based on parent/guardian self-report of child's condition and responses to category M on the CASI-5 subscale.
* Any serious medical condition, including inflammatory bowel disease, history of cancer, kidney or liver disease, hyperthyroidism, diabetes Type I or II.
* Known allergy to any ingredients of the intervention.
* Any known abnormality of mineral metabolism (e.g., Wilson's disease, hemochromatosis).
* Taking any other medication with primarily central nervous system activity, including stimulants, within the last two weeks prior to in-person assessment; participants must be off these medications for a minimum of two weeks prior to the screening.
* Severe separation anxiety that would preclude separating from parent/guardian to answer study questionnaires.
* Any disability that would interfere with participant answering questions verbally.
* Non-English speaking.
* Pregnancy or sexually active at baseline. Exclusion criteria 1-6 and 9, will be based on parent/guardian self-report of child's condition. If the parent/guardian reports medical exclusion criteria, or concerns about eligibility, data provided by parent/guardian will be confirmed by review of medical records with release of information signed by parent/guardian. Potential participant may be reviewed in-person by a study physician in the case of any concerns about participation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Johnstone, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
- University of Lethbridge, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robinette LM, Hatsu IE, Adetona O, Wu CM, Johnstone JM, Bruton AM, Ast HK, Odei JB, Ziouzenkova O, Leung BMY, Arnold LE. Multinutrients Decrease Oxidative Stress in Children With ADHD: Mediation/Moderation Analysis of Randomized Controlled Trial Data. J Atten Disord. 2025 Dec;29(14):1290-1306. doi: 10.1177/10870547251355998. Epub 2025 Aug 7. PMID 40772654
- [Derived] Leung BMY, Srikanth P, Gracious B, Hatsu IE, Tost G, Conrad V, Johnstone JM, Arnold LE. Paediatric adverse event rating scale: a measure of safety or efficacy? Novel analysis from the MADDY study. Curr Med Res Opin. 2022 Sep;38(9):1595-1602. doi: 10.1080/03007995.2022.2096333. Epub 2022 Jul 11. PMID 35770861
- [Derived] Johnstone JM, Hatsu I, Tost G, Srikanth P, Eiterman LP, Bruton AM, Ast HK, Robinette LM, Stern MM, Millington EG, Gracious BL, Hughes AJ, Leung BMY, Arnold LE. Micronutrients for Attention-Deficit/Hyperactivity Disorder in Youths: A Placebo-Controlled Randomized Clinical Trial. J Am Acad Child Adolesc Psychiatry. 2022 May;61(5):647-661. doi: 10.1016/j.jaac.2021.07.005. Epub 2021 Jul 22. PMID 34303786
- [Derived] Johnstone JM, Leung B, Gracious B, Perez L, Tost G, Savoy A, Hatsu I, Hughes A, Bruton A, Arnold LE. Rationale and design of an international randomized placebo-controlled trial of a 36-ingredient micronutrient supplement for children with ADHD and irritable mood: The Micronutrients for ADHD in Youth (MADDY) study. Contemp Clin Trials Commun. 2019 Oct 26;16:100478. doi: 10.1016/j.conctc.2019.100478. eCollection 2019 Dec. PMID 31763491

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: Intervention & Placebo
Arm/Group | Intervention | Placebo | Open Label
Started | 78 | 57 | 0
Completed | 69 | 54 | 0
Not Completed | 9 | 3 | 0
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Unable to swallow pills | 4 | 1 | 0
Not completed — Commenced stimulant medication | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Period: Phase 2: Open Label
Arm/Group | Intervention | Placebo | Open Label
Started | 0 | 0 | 123
Completed | 0 | 0 | 99
Not Completed | 0 | 0 | 24
Not completed — Commenced stimulant medication | 0 | 0 | 3
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 78 | 57 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 78 | 57 | 135
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 57 | 35 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — "Other" ethnicity includes Jewish, Japanese, European, Metis, Canadian, or other/not specified
  Participants
    Ethnicity: Not Hispanic or Latino | 45 | 40 | 85
    Ethnicity: Hispanic or Latino | 7 | 1 | 8
    Ethnicity: Other | 4 | 3 | 7
    Ethnicity: Unknown/Did Not Report | 22 | 13 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — "Other" includes American Indian/Native American or Alaska Native, Metis, Native Hawaiian/Pacific Islander, or not specified.
  Participants
    Race: Asian | 3 | 0 | 3
    Race: African American/Black | 1 | 3 | 4
    Race: White | 60 | 45 | 105
    Race: Other | 3 | 4 | 7
    Race: Unknown/Not Reported | 11 | 5 | 16
Region of Enrollment [Number; unit: participants] — Population: Participants included in the ITT analysis.
  participants
    Canada: number analyzed (Participants) | 71 | 55 | 126
    Canada | 21 | 17 | 38
    United States: number analyzed (Participants) | 71 | 55 | 126
    United States | 50 | 38 | 88

OUTCOME MEASURES:

1. Primary Outcome: CASI-5 Parent-rated Composite Score
Description: Primary outcome measure, defined a priori, reflecting the often-comorbid ADHD symptoms of emotional dysregulation irritable mood, anger or aggression), are the parent-rated Child and Adolescent Symptom Inventory (CASI-5). The CASI-5 is based on the DSM-5 symptom criteria. The subscales of ADHD, Oppositional Defiant Disorder (ODD), Disruptive Mood Dysregulation Disorder (DMDD) and peer conflict that will be combined into a total composite score; range is 0-3 (never, sometimes, often, very often). Higher scores represent a worse outcome.
Time Frame: Baseline and week 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 78 | 57
score on a scale
  Baseline | 1.49 (0.08) | 1.52 (0.08)
  Week 8 | 1.18 (0.08) | 1.23 (0.08)

2. Primary Outcome: Clinical Global Impression (CGI) - Number of Participants Considered a Treatment Responder (Score of 1 or 2)
Description: Second primary measure is the blinded clinician-rated CGI-Improvement (CGI-I) is a subscale of the CGI that rates overall improvement of symptoms based on all relevant data. Item range is 1-7 (very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse); lower score is better. A treatment responder is defined as a participant who is rated a 1 or 2 on the CGI-I. The CGI-Severity (CGI-S) subscale will also be scored at baseline and week 8, with scores compared at the two time points. Item range is 1-7 (normal, borderline ill, mildly ill, moderately ill, markedly ill, severely ill, among the most extremely ill patients); lower score is better; most participants will be a 4 or 5 at baseline.
Time Frame: Week 8
Population: Participants considered in the ITT analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 71 | 55
Participants | 38 | 10

3. Secondary Outcome: Sodium, Potassium, Chloride, Carbon Dioxide, and Anion Gap in mmol/L
Description: Collect blood and urine samples at two time points. The samples are being collected per a request from the FDA for safety screening.
Time Frame: Baseline and Week 8
Population: Only participants in the US sites provided blood and urine samples. Canadian participants were not required by Health Canada to collect safety blood or urine samples, hence the lower number of participants.
Measure: Mean (Standard Error); unit: mmol/L
Groups:
- Intervention (Baseline); Intervention (Week 8): Capsules of broad spectrum micronutrients: a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants.
  Broad Spectrum Micronutrients; a 36-ingredient blend of vitamins, minerals, amino acids, and antioxidants: 60% of participants will take 3-4 capsules of broad spectrum micronutrients three times per day for eight weeks. Following the initial 8 weeks (of the RCT), all participants will have the option to participate in an open label extension, during which time the child would take the active micronutrient treatment for 8 weeks
- Placebo (Baseline); Placebo (Week 8): Capsules of inactive placebo.
  Placebo: 40% of participants will take 3-4 capsules of inactive placebo three times per day for eight weeks.
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
mmol/L
  Sodium | 139.13 (0.34) | 139.16 (0.34) | 139.28 (0.36) | 139.42 (0.37)
  Potassium | 4.1 (0.10) | 4.06 (0.10) | 4.09 (0.10) | 4.0 (0.10)
  Chloride | 105.07 (0.96) | 104.81 (0.97) | 104.88 (0.97) | 105.28 (0.98)
  Carbon dioxide | 25.62 (0.21) | 25.64 (0.22) | 25.97 (0.24) | 25.86 (0.25)
  Anion gap | 10.30 (2.83) | 10.64 (2.83) | 10.31 (2.83) | 10.15 (2.84)

4. Secondary Outcome: Calcium, Blood Urea Nitrogen, Creatinine, Glucose, Bilirubin Total in mg/dL
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
mg/dL
  Calcium | 9.47 (0.20) | 9.49 (0.20) | 9.47 (0.20) | 9.40 (0.20)
  Blood urea nitrogen (BUN) | 12.48 (0.41) | 13.17 (0.42) | 12.56 (0.46) | 12.13 (0.48)
  Creatinine | 0.46 (0.01) | 0.49 (0.01) | 0.46 (0.01) | 0.46 (0.01)
  Glucose | 82.15 (2.36) | 83.03 (2.39) | 79.45 (2.44) | 80.0 (2.46)
  Bilirubin total | 0.47 (0.03) | 0.45 (0.03) | 0.49 (0.03) | 0.46 (0.03)

5. Secondary Outcome: Albumin, Total Protein, Hemoglobin, Mean Cell Hgb in g/dL
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
g/dL
  Albumin | 4.34 (0.17) | 4.34 (0.17) | 4.29 (0.17) | 4.28 (0.17)
  Total protein | 7.15 (0.63) | 8.45 (0.65) | 7.07 (0.73) | 7.06 (0.76)
  Hemoglobin | 12.99 (0.17) | 12.96 (0.17) | 12.99 (0.18) | 12.91 (0.18)
  Mean cell Hgb concentration | 33.82 (0.13) | 33.59 (0.13) | 33.75 (0.15) | 33.47 (0.15)

6. Secondary Outcome: AST, ALT, Alkaline in U/L
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
U/L
  AST | 23.58 (1.26) | 27.28 (1.28) | 25.72 (1.42) | 22.79 (1.46)
  ALT | 18.67 (3.25) | 26.00 (3.27) | 20.40 (3.37) | 18.09 (3.41)
  Alkaline phosphatase | 255 (8.10) | 241.33 (8.15) | 252.21 (9.29) | 257.93 (9.41)

7. Secondary Outcome: RBC Count in Cells/mcL
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cells/mcL
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
cells/mcL | 4,650,000 (0.08) | 4,650,000 (0.08) | 4,600,000 (0.08) | 4,600,000 (0.09)

8. Secondary Outcome: Hematocrit, RBC Distribution, Immature Grans, Lymphocyte, Monocyte, Eosinophil in Percent
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percent
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
percent
  Hematocrit | 38.40 (0.52) | 38.60 (0.52) | 38.50 (0.55) | 38.60 (0.55)
  RBC distribution | 25.03 (8.76) | 25.17 (8.76) | 25.29 (8.76) | 25.02 (8.76)
  Immature grans | 0.20 (0.02) | 0.18 (0.02) | 0.24 (0.02) | 0.19 (0.03)
  Lymphocyte | 43.63 (1.65) | 43.53 (1.66) | 40.25 (1.80) | 40.65 (1.84)
  Monocyte | 8.03 (0.34) | 8.29 (0.34) | 7.78 (0.38) | 8.35 (0.38)
  Eosinophil | 3.82 (0.63) | 4.03 (0.64) | 6.49 (0.73) | 5.71 (0.75)

9. Secondary Outcome: Mean Cell Volume in fL
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: fL
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
fL | 82.70 (0.44) | 83.00 (0.45) | 83.74 (0.49) | 83.85 (0.50)

10. Secondary Outcome: Iron in ug/dL
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: ug/dL
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
ug/dL | 99.1 (4.65) | 90.7 (4.69) | 100.5 (5.35) | 95.5 (5.49)

11. Secondary Outcome: WBC Count, Absolute Monocyte, Absolute Eosinophil, Platelet Count in Cells/mcL
Description: as for outcome 3
Time Frame: Baseline and Week 8
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cells/mcL
Arm/Group | Intervention (Baseline) | Intervention (Week 8) | Placebo (Baseline) | Placebo (Week 8)
Number analyzed (Participants) | 50 | 50 | 38 | 38
cells/mcL
  WBC count | 5,710 (0.22) | 5,730 (0.23) | 6,080 (0.25) | 5,990 (0.26)
  Absolute monocyte | 460 (0.02) | 470 (0.02) | 460 (0.02) | 480 (0.02)
  Absolute eosinophil | 210 (0.04) | 230 (0.04) | 390 (0.04) | 340 (0.05)
  Platelet count | 289,970 (7.54) | 289,320 (7.57) | 290,160 (8.62) | 295,900 (8.75)

12. Secondary Outcome: Clinical Global Impression (CGI)
Description: as for outcome 2
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Open Label (Week 8 to Week 16): All children knowingly received the active intervention
Arm/Group | Open Label (Week 8 to Week 16)
Number analyzed (Participants) | 103
Participants | 103

13. Secondary Outcome: CASI-5 Parent Report
Description: Primary outcome measure, defined a priori, reflecting the often-comorbid ADHD symptoms of emotional dysregulation irritable mood, anger or aggression), are the parent-rated Child and Adolescent Symptom Inventory (CASI-5) subscales of ADHD, Oppositional Defiant Disorder (ODD), Disruptive Mood Dysregulation Disorder (DMDD) and peer conflict. The CASI-5 is based on the DSM-5 symptom criteria. Item range is 0-3 (never, sometimes, often, very often). Higher scores represent a worse outcome. The subscales for ADHD, ODD, and DMD will be composite scores.
Time Frame: Week 16
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Open Label (Week 8 to Week 16)
Number analyzed (Participants) | 103
score on a scale
  Week 12 | 1.14 (0.04)
  Week 16 | 0.99 (0.05)

ADVERSE EVENTS:
Time Frame: Baseline, week 1, week 4, week 8 and week 16
Description: Used the Pediatric Adverse Events Rating Scale (PAERS) to assess treatment emergent adverse events.
Arm/Group | Intervention | Placebo | Open Label
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/54 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/54 | 0/99
Other Adverse Events (participants affected / at risk) | 22/69 | 24/54 | 26/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=69) | Placebo (N=54) | Open Label (N=99)
Irritability (Psychiatric disorders) | 1 | 1 | 0
Angry or hostile (Psychiatric disorders) | 3 | 1 | 2
Sad or low mood (Psychiatric disorders) | 2 | 0 | 3
Lack of interest (Psychiatric disorders) | 2 | 0 | 1
Mood swings (Psychiatric disorders) | 2 | 1 | 2
Anxious, tense, or uptight (Psychiatric disorders) | 3 | 1 | 2
Lack of self-control/ impulsive (Psychiatric disorders) | 3 | 2 | 1
Trouble paying attention or concentrating (Psychiatric disorders) | 2 | 0 | 0
Racing thoughts (Psychiatric disorders) | 1 | 1 | 0
Can't sit or stand still (Psychiatric disorders) | 3 | 1 | 0
Tired/fatigued (General disorders) | 2 | 1 | 0
Trouble falling asleep (General disorders) | 4 | 1 | 0
Tried to hurt himself/ herself (Psychiatric disorders) | 1 | 0 | 1
Hurt someone or something (Psychiatric disorders) | 1 | 1 | 1
Less hungry (Metabolism and nutrition disorders) | 4 | 1 | 4
Lost weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Dry mouth (Metabolism and nutrition disorders) | 1 | 0 | 0
Gained weight (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle shaking, stiffness, or cramps (Nervous system disorders) | 0 | 1 | 0
Tics (Nervous system disorders) | 0 | 1 | 0
Unusually good mood or super happy (Psychiatric disorders) | 1 | 1 | 2
Skin rash or irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Heart racing or skipping beats (Cardiac disorders) | 0 | 1 | 0
GI symptoms (Gastrointestinal disorders) | 17 | 8 | 9 — GI symptoms are a combination of discrete participants experiencing stomach ache or cramps, nausea/sick to stomach, throwing up/vomiting, and diarrhea.
Headache (Nervous system disorders) | 1 | 2 | 0
Other (General disorders) | 5 | 5 | 2
Chest Pain (General disorders) | 0 | 0 | 1
Dizzy or light-headed (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03252522/Prot_SAP_001.pdf